CLINICAL TRIAL: NCT01449422
Title: Evaluation Of The Efficacy, Tolerance And Acceptability Of URGO Dressing 310 3082 Versus A Hydrofibre Dressing In The Local Management Of Venous Or Predominantly Venous Mixed Leg Ulcers
Brief Title: Clinical Trial to Evaluate the Efficacy, Tolerance and Acceptability of URGO Dressing vs a Hydrofibre in the Local Management of Venous or Predominantly Venous Mixed Leg Ulcers.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoires URGO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FI-11-02-310 3082
Record Dates: First submitted 2011-10-03; First posted 2011-10-10 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Varicose Ulcer
MeSH Terms: conditions — Varicose Ulcer | interventions — Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- URGO 310 3082 (Experimental)
  Interventions: Device: Dressing
- Aquacel (Active Comparator)
  Interventions: Device: Dressing

INTERVENTIONS:
Device: Dressing — the dressing should be changed on average every 1 to 2 days, then as often as required (up to 7 days) depending on the exudate volume and the clinical condition of the wound (evaluated by the investigating doctor).
  Arms: URGO 310 3082
Device: Dressing — the hydrofibre dressing should be changed when it is saturated, or depending on the clinical appreciation of the situation. The dressing can remain in place for up to 7 days.
  Arms: Aquacel

SUMMARY:
The main objective of this trial is to demonstrate that a local care strategy using URGO 310 3082 dressing is not inferior to a reference therapeutic strategy using a hydrofibre dressing in the management of venous ulcers. This non-inferiority hypothesis will be judged on the planimetric relative regression of the wound surface area after six weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old who has provided his/her written informed consent
* Patient who can be monitored by the same investigation team throughout the duration of the study
* Patient who agrees to wear effective venous compression every day, associated with the trial dressing
* Leg ulcer with a distal Ankle Brachial Pressure Index (ABPI) not less than 0.7 and not more than 1.3
* Ulcer with a minimum area of 3 cm2 and a maximum area of 30 cm2
* Ulcer duration between 3 and 36 months
* Ulcer where the surface area is 70% or more covered by fibrinous tissue
* Ulcer at least 3 cm away from any other lesion
* Ulcer moderately or strongly exudative justifying the use of an absorbent dressing

Exclusion Criteria:

* Female patient of child-bearing potential who has no effective means of contraception
* Patient who is pregnant or breastfeeding
* Patient taking part in another therapeutic trial
* Patient with hypersensitivity to one of the components of the trial dressing or a known allergy to carboxymethylcellulose (hydrocolloid)
* Patient with a serious general pathological condition who, it may be feared, might discontinue participation in the trial before the six weeks of treatment
* Patient with an evolving neoplastic condition, treated by radiotherapy, chemotherapy or hormone therapy
* Patient with a systemic infection not controlled by suitable antibiotic treatment
* Patient who, during the 3 months before inclusion, presented a deep vein thrombosis
* Ulcer where its surface is totally or partially covered by black necrotic plaque
* Ulcer which is clinically infected
* Ulcer requiring surgical treatment or for which surgery is programmed during the six weeks following inclusion
* Malignant ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The efficacy of dressings under trial will be judged on the evolution of wound surface area after six weeks of treatment. | Week 1, 2, 4 and 6
  The main evaluation criterion is the relative planimetric regression of the wound surface area, calculated according to the following formula, from centralised planimetric measurements:
  Regression of the area (%) = [(ST0-STlast)/ST0] x 100 ST0: Surface area of the lesion measured on the day of inclusion STlast: Surface area of the lesion at the last planimetric evaluation available

SECONDARY OUTCOMES:
Comparison between the two devices of percentage of lesions in which the evolution is positive (defined by a relative regression at least 40% of wound surface) after monitoring for 6 weeks. | Week 1, 2, 4 and 6
Comparison between the two groups of percentage of debrided lesions (defined by a lesion with more than 70% of its surface covered by granulation tissue of a "red colour" on the colorimetric scale), at the last available evaluation | Week 1, 2, 4 and 6
Comparison between the two strategies of percentage of patients in whom at least one problem of pain was detected during care (VAS score at the end of care > 30 mm) | Week 1, 2, 4 and 6
Comparison between the 2 groups of the percentage of wound care associated with manual debridement | Week 1, 2, 4 and 6
Comparison between the two groups of the evolution of the patients' quality of life between inclusion and the last available visit. This quality of life will be assessed using the EuroQol-5D™ questionnaire | Week 1, 2, 4 and 6
Comparison between the 2 groups of the percentage of the participants number with Adverse Events | Week 1, 2, 4 and 6
Comparison between the 2 groups of the mean number of dressing changes per week. | Week 1, 2, 4 and 6
Comparison between the 2 groups of the easiness application and removal | Week 1, 2, 4 and 6
Comparison between the 2 groups of the percentage of good or very good conformability | Week 1, 2, 4 and 6
Comparison between the 2 groups of the mean value for overall performance score | Week 1, 2, 4 and 6
  This score will be between 0 and 36

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Rothschild, Paris, France